CLINICAL TRIAL: NCT05449561
Title: Beyond Efficacy- Eliciting Preference for Face-to-face and Internet-based Psychotherapy Among People with Depression: Using Discrete Choice Experiment to Advance Future Service Implementation
Brief Title: Beyond Efficacy- Eliciting Preference for Face-to-face and Internet-based Psychotherapy Among People with Depression
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Winnie W.S. MAK, Professor, Chinese University of Hong Kong
Other Study IDs: SBRE(R)-21-043
Record Dates: First submitted 2022-06-29; First posted 2022-07-08 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Depression
Keywords: mental well-being; depression; Internet-based Psychotherapy; Client-Centered Services; Discrete Choice Experiment (DCE)
MeSH Terms: conditions — Depression; Psychological Well-Being

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Discrete Choice qualitative interview: We will invite at least 20 participants with at least mild level of depressive symptoms to participate in individual interviews. The interviews will be in semi-structured format. Upon provision of informed consent and completion of demographics survey, we will ask respondents a single question of what matters to them when considering the use of psychotherapy, with adequate probes during the conversation. This will ensure uniformity of the topics to be discussed, and the level of digression allowed.

SUMMARY:
The aim of this study is to strengthen the evidence base of clients' preferences of psychotherapy and to close the described literature gaps so as to inform public health resource reallocation and implementation of psychological services.

The investigators aim to address the following research questions:

1. Which psychological service attributes exert the most inﬂuence on the service use decisions?
2. Can respondents be represented by latent classes on the basis of similar preference profiles?
3. Which attributes exert the most inﬂuence on the service utilization decisions of each latent class?
4. Will people with depression adopt Internet-based psychotherapy considering the long waiting time and high cost of conventional face-to-face psychotherapy?

To systematically address the above questions, specific research objectives are defined as follows:

1. to examine the relative importance of a series of characteristics of psychological services (e.g., delivery modality, waiting time, out-of-pocket service fee, anonymity and referral methods) on the choices of psychological service using DCE.
2. to identify segments of people with depression with different service preferences using latent class model, because the relative weighting of service preferences may vary with demographic (e.g., gender, age, socioeconomic status, depression severity) and psychological characteristics (e.g., help seeking stigma); and
3. since DCEs need to be translated into improved services to be truly useful, and with reference to emerging interest in the development of digital mental health service for people with depression to solve the issue of long waiting time and cost in face-to-face psychotherapy, using a series of statistical simulations, we aim to estimate the percentage of people with depression in each latent class segment who would use psychotherapy with pre-defined treatment attributes packages.

DETAILED DESCRIPTION:
1.1 Depression and Internet-based Psychotherapy as a way to improve Access of Care Depression is a common mental disorder with a prevalence of 8.8%. It is associated with a significant decrement of quality of life, ranked as the 3rd cause of burden of disease worldwide by WHO and will be ranked 1st by 2030(1). Nonetheless, 55.3% people with depression were unwilling to seek professional help for depression(2), and the median duration of delay in treatment ranges from 2 to 8 years(3,4). Although a preference for psychotherapy over pharmacological treatment was consistently evident(5), barriers to traditional face-to-face psychotherapy such as inconvenient location, long waiting time, high costs, low perceived need, preference to self-reliance, self-stigma, and feelings of embarrassment (6) deter many to access and adhere to treatment. Worse still, the number of individuals with mental disorders has far outnumbered the resources available in traditional models of delivering psychotherapy(7). Thus, effective psychotherapies need to be made increasingly available in a more cost-effective way using the Internet as an alternative service modality(8). Research suggests that the less labor-intensive Internet-based psychotherapies appear to be an effective strategy in increasing psychosocial services and reducing burden to the healthcare system. Numerous clinical trials have demonstrated the efficacy of Internet-based psychotherapies in treating depression. A systematic review of 32 randomized controlled trials evaluating Internet-based cognitive behavioral therapy for symptoms of depression in 5642 participants found a mean effect size of g=0.67 (8). A recent meta-analysis also found that Internet-based cognitive behavioral psychotherapy has comparable effects to traditional face-to-face psychotherapy, even when they are compared directly to each other(9).

1.2 Beyond Efficacy, the Importance of Preference in Client-Centered Services Despite the growing evidence on the equivalence of efficacy in using the Internet to deliver psychotherapy as compared to its face-to-face counterpart, an essential prerequisite to actualize the full potential of any effective treatment is that individuals are willing to utilize it. This proposition is in accordance with the Diffusion of Innovation Theory and The Unified Theory of Acceptance and Use of Technology; potential users need to have an adequate level of service preference and acceptance prior to the initiation and uptake of the novel treatment(10).With the awareness of translational issues (e.g., poor uptake) occurring from efficacy trials to the real world and the recognition that healthcare interventions are valued for more than just clinical health outcomes(11), research in understanding what patients* care in health services had a ten-fold increase in the last two decades(12). In fact, involving patients' preferences in the determination of best care not only leads to better service implementation, it also promote policy decisions that embrace patient values(13). Unmet preferences partly explain the sub-optimal uptake and poor adherence of psychotherapy for major depressive disorder(14,15). Addressing client preferences for psychotherapies could help overcome the treatment gap by guiding policy decisions and restructuring psychological services offered in the society(11). Characterizing and prioritizing potential service users' demand for evidence-based psychotherapies could provide insights to such significant and practical questions as "To whom should Internet-based psychotherapy be implemented?", "How should resources be allocated between Internet-based and face-to-face services to commensurate with users' preferences?" "Can the new service modality reach people who have high levels of stigma or prefer managing their mental health anonymously through an online program?(16)". Unsurprisingly, research found that accounting for patients' preference in service planning could lead to improved service utilization and decreased dropout(17). The UK National Health Services also explicitly stated its "services must reflect, and should be coordinated around and tailored to, the needs and preferences of patients". Furthermore, respect of users' autonomy and self-determination is recognized in international Code of Ethics including those of the American and the Australian Psychological Society. Patients' preference was also identified as one of the six aims for high-quality new health system for the 21st century in the Institute of Medicine report, Crossing the Quality Chasm.

1.3 Using Discrete Choice Experiment (DCE) to understand client preferences To date, client preferences in psychological services have primarily been assessed using qualitative methods or quantitative measures of acceptability or attitudes(18). Studies suggested the mean preference strength of Internet-based psychotherapy was lower than traditional psychotherapy, yet comparable to that of medication. A substantial portion of people with depression (38%) reported likely or very likely to consider Internet-based interventions (18). For those preferring traditional face-to-face approaches, more than a third of them indicated that they are likely to use online services in the future(19). In a recent preference study in Canada, although most postsecondary students preferred face-to-face psychotherapy over the digital mental health service, when students considered potential waiting periods, a greater percentage of students opted for Internet-based psychotherapy over waiting for face-to-face psychotherapy (20). Although preference studies using simple Likert scale ratings provided certain insight into desirable service, they lacked details on the underlying attributes that drive user preferences, and they did not quantitatively assess the relative importance of each attribute (e.g., 'Is the treatment modality, waiting duration, or cost the most important?') or the degree to which clients would be willing to trade-oﬀ one treatment characteristic for another (e.g., 'Would clients be willing to receive services via the Internet as opposed to in-person if it reduces cost/waiting time?'). Without this information, researchers and policy makers have limited guidance on how best to design best services that align with client preferences.

An alternative to preference studies is discrete choice experiment (DCE), which can be used to quantitatively, experimentally and systematically understand clients' preference. DCE is a valid, reliable, and widely applied survey methodology for eliciting patients' preferences for health care(21). DCE is grounded in random utility theory that posits individuals choosing attributes that maximize the option utility. In DCE, respondents will be asked to complete a series of hypothetical choice tasks (see Figure 2 for example). Within each task, the respondents select their preferred option from alternatives with varying service characteristics. DCE is analogous to real-world decision making and offer advantages over traditional survey methods in reducing superficial decision-making, halo effect and social desirability bias, and allowing a better understanding of the underlying reasons of choice behaviors(22). Ratings often produce high scores across favorable attributes, reﬂecting general desire for services that encompass all positive characteristics. However, the scarcity of resources often necessitates trade-offs between attributes, and DCE could provide important information to inform services decision making on what service attributes are to be prioritized for improvement(21). Notably, DCE is simple to administer, with studies showing individuals with severe mental illnesses capable of completing DCE and making rational decisions (23), and choice methods has been found to adequately predict actual behavior(24).

In fact, the United States Food and Drug Administration has endorsed DCEs as the 'favored' method for assessing patients view on harm and benefit profile of health care products. Similarly, data derived from DCEs also played a signiﬁcant role in informing and supporting health care decision making and regulation(25). In the field of academia, researchers have applied DCEs to identify attributes that impact patient preferences for breast cancer screening programs (26), HIV prevention (27), rheumatoid arthritis treatment(28), and vaccination(24). Given DCE can capture the relative importance of the studied attributes, intervention researchers and policy makers can prioritize the changes related to the most important attribute in psychotherapy in service development and implementation.

1.4 The Research Gap: What about relative significance of important service attributes? Hitherto, only a handful of DCEs have been conducted on psychological services. Prioritizing services on the basis of clinical efficacy and cost-effectiveness often overlooks other important factors relevant to the clients. Capturing clients' choices in psychotherapy in light of the new development in Internet-based interventions is of paramount importance and urgency to optimize service implementation(11).

To the best of our knowledge, only one study to date has explicitly examined how people with depression trade off the pros and cons of psychological service options with varying service attributes(29). However, the study adopted forced choice tasks without an opt-out alternative, making choice sets less realistic and at risk of preference weight over-estimation (30,31). Moreover, no existing DCE on psychological services has incorporated all the three main treatment attributes for depression, which are outcome (e.g., effectiveness), process (e.g., treatment modality, waiting time), and cost attributes(32) 1.5 Study Aim The aim of this study is to strengthen the evidence base of clients' preferences of psychotherapy and to close the described literature gaps so as to inform public health resource reallocation and implementation of psychological services. The investigators aim to address the following research questions: ‣ Which psychological service attributes exert the most inﬂuence on the service use decisions? ‣ Can respondents be represented by latent classes on the basis of similar preference profiles? Which attributes exert the most inﬂuence on the service utilization decisions of each latent class? ‣ Will people with depression adopt Internet-based psychotherapy considering the long waiting time and high cost of conventional face-to-face psychotherapy?

To systematically address the above questions, specific research objectives are defined as follow:

1. to examine the relative importance of a series of characteristics of psychological services (e.g., delivery modality, waiting time, out-of-pocket service fee, anonymity and referral methods) on the choices of psychological service using DCE.
2. to identify segments of people with depression with different service preferences using latent class model, because the relative weighting of service preferences may vary with demographic (e.g., gender, age, socioeconomic status, depression severity) and psychological characteristics (e.g., help seeking stigma); and
3. since DCEs need to be translated into improved services to be truly useful, and with reference to emerging interest in the development of digital mental health service for people with depression to solve the issue of long waiting time and cost in face-to-face psychotherapy, using a series of statistical simulations, the investigators aim to estimate the percentage of people with depression in each latent class segment who would use psychotherapy with pre-defined treatment attributes packages.

Afterwards, the investigators will invite at least 20 participants with at least mild level of depressive symptoms to participate in individual interviews. The interviews will be in semi-structured format.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 years old or above
* With at least mild to moderate depressive symptoms (defined as having a cut-off score of 10 or above based on the Patient Health Questionnaire-9 (PHQ-9))
* Able to read and understand Chinese

Exclusion Criteria:

* Self-reported DSM-5 diagnosis of current manic episodes, post-traumatic stress disorder, substance use disorders, and psychotic disorders
* Actively suicidal as assessed by P4-suicidality screener

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A variety of online and offline approaches to recruit a diverse sample of people with depression. Participants will be recruited using both online and offline approaches, including social/digital media and print media advertisement, forums, mutual support groups for people with depression, Integrated Community Centers for Mental Wellness, primary health clinics. Quota sampling on gender, age, and socioeconomic status will be adopted. The inclusion criteria include: (1) aged 18 years old or above (2) with at least mild to moderate depressive symptoms (defined as having a cut-off score of 10 or above based on the Patient Health Questionnaire-9 (PHQ-9)) (3) able to read and understand Chinese. Exclusion criteria include: (1) self-reported DSM-5 diagnosis of current manic episodes, post-traumatic stress disorder, substance use disorders, and psychotic disorders (2) actively suicidal as assessed by P4-suicidality screener.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
Depression | at baseline
  Patient Health Questionnaire (PHQ9) (Kroenke, Spitzer, & Williams, 2001). It is a 9-item measure to access the severity of depression. PHQ-9 has been validated and used widely in the general population for screening and measuring depression severity. Scores of 5, 10, 15, and 20 denote mild, moderate, moderately severe, and severe level of depression respectively (range: 0-27).
Help-seeking Self-Stigma | at baseline
  Self-Stigma of Seeking Help Scale (SSOSH-10). To understand how stigma may influence choices and preference of psychological service, SSOSH-10 will be used to assess respondents' level of help seeking stigma. The scale scores on a 5-point Likert-type scale, with 1= totally disagree and 5 = totally agree (scores range from 10 to 50). The higher the mean score, the higher the self-stigma of seeking help.
Attitudes towards Psychological Online Interventions | at baseline
  Attitudes towards Psychological Online Interventions Questionnaire (APOI). It is a 16-item measure to assess respondent's attitudes towards psychological online interventions. It scores on a 5-point Likert scale with 1=totally agree to 5=totally disagree.
Potential attributes and their influence on respondent's choice of psychotherapies | baseline (During qualitative interview)
  1 set of questions with different attributes that influence respondent's choice of psychotherapy will be asked. We plan to include (1) Treatment Modality, (2) Effectiveness, (3) Referral, (4) Anonymity, (5) Waiting Time and (6) Out-Of-Pocket Cost as attributes. We will also ask another 60 participants with depressive symptoms to rank attributes from 1 ("most important") to 9 ("least important"). The 6 highest ranked attributes will be selected for the questions.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychology, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Malhi GS, Mann JJ. Depression. Lancet. 2018 Nov 24;392(10161):2299-2312. doi: 10.1016/S0140-6736(18)31948-2. Epub 2018 Nov 2. PMID 30396512
- [Background] Yoshikawa E, Taniguchi T, Nakamura-Taira N, Ishiguro S, Matsumura H. Factors associated with unwillingness to seek professional help for depression: a web-based survey. BMC Res Notes. 2017 Dec 4;10(1):673. doi: 10.1186/s13104-017-3010-1. PMID 29202791
- [Background] Stagnaro JC, Cia AH, Vommaro H, Sustas S, Vazquez N, Serfaty E, Kessler RC, Benjet C. Delays in making initial treatment contact after the first onset of mental health disorders in the Argentinean Study of Mental Health Epidemiology. Epidemiol Psychiatr Sci. 2019 Apr;28(2):240-250. doi: 10.1017/S2045796018000094. Epub 2018 Mar 15. PMID 29540248
- [Background] Wang PS, Angermeyer M, Borges G, Bruffaerts R, Tat Chiu W, DE Girolamo G, Fayyad J, Gureje O, Haro JM, Huang Y, Kessler RC, Kovess V, Levinson D, Nakane Y, Oakley Brown MA, Ormel JH, Posada-Villa J, Aguilar-Gaxiola S, Alonso J, Lee S, Heeringa S, Pennell BE, Chatterji S, Ustun TB. Delay and failure in treatment seeking after first onset of mental disorders in the World Health Organization's World Mental Health Survey Initiative. World Psychiatry. 2007 Oct;6(3):177-85. PMID 18188443
- [Background] McHugh RK, Whitton SW, Peckham AD, Welge JA, Otto MW. Patient preference for psychological vs pharmacologic treatment of psychiatric disorders: a meta-analytic review. J Clin Psychiatry. 2013 Jun;74(6):595-602. doi: 10.4088/JCP.12r07757. PMID 23842011
- [Background] Andrade LH, Alonso J, Mneimneh Z, Wells JE, Al-Hamzawi A, Borges G, Bromet E, Bruffaerts R, de Girolamo G, de Graaf R, Florescu S, Gureje O, Hinkov HR, Hu C, Huang Y, Hwang I, Jin R, Karam EG, Kovess-Masfety V, Levinson D, Matschinger H, O'Neill S, Posada-Villa J, Sagar R, Sampson NA, Sasu C, Stein DJ, Takeshima T, Viana MC, Xavier M, Kessler RC. Barriers to mental health treatment: results from the WHO World Mental Health surveys. Psychol Med. 2014 Apr;44(6):1303-17. doi: 10.1017/S0033291713001943. Epub 2013 Aug 9. PMID 23931656
- [Background] Kazdin AE, Blase SL. Rebooting Psychotherapy Research and Practice to Reduce the Burden of Mental Illness. Perspect Psychol Sci. 2011 Jan;6(1):21-37. doi: 10.1177/1745691610393527. Epub 2011 Feb 3. PMID 26162113
- [Background] Andrews G, Basu A, Cuijpers P, Craske MG, McEvoy P, English CL, Newby JM. Computer therapy for the anxiety and depression disorders is effective, acceptable and practical health care: An updated meta-analysis. J Anxiety Disord. 2018 Apr;55:70-78. doi: 10.1016/j.janxdis.2018.01.001. Epub 2018 Feb 1. PMID 29422409
- [Background] Andersson G, Topooco N, Havik O, Nordgreen T. Internet-supported versus face-to-face cognitive behavior therapy for depression. Expert Rev Neurother. 2016;16(1):55-60. doi: 10.1586/14737175.2015.1125783. Epub 2015 Dec 15. PMID 26610160
- [Background] Musiat P, Goldstone P, Tarrier N. Understanding the acceptability of e-mental health--attitudes and expectations towards computerised self-help treatments for mental health problems. BMC Psychiatry. 2014 Apr 11;14:109. doi: 10.1186/1471-244X-14-109. PMID 24725765
- [Background] Salloum RG, Shenkman EA, Louviere JJ, Chambers DA. Application of discrete choice experiments to enhance stakeholder engagement as a strategy for advancing implementation: a systematic review. Implement Sci. 2017 Nov 23;12(1):140. doi: 10.1186/s13012-017-0675-8. PMID 29169397
- [Background] Clark MD, Determann D, Petrou S, Moro D, de Bekker-Grob EW. Discrete choice experiments in health economics: a review of the literature. Pharmacoeconomics. 2014 Sep;32(9):883-902. doi: 10.1007/s40273-014-0170-x. PMID 25005924
- [Background] Bridges JF, Hauber AB, Marshall D, Lloyd A, Prosser LA, Regier DA, Johnson FR, Mauskopf J. Conjoint analysis applications in health--a checklist: a report of the ISPOR Good Research Practices for Conjoint Analysis Task Force. Value Health. 2011 Jun;14(4):403-13. doi: 10.1016/j.jval.2010.11.013. Epub 2011 Apr 22. PMID 21669364
- [Background] Renn BN, Hoeft TJ, Lee HS, Bauer AM, Arean PA. Preference for in-person psychotherapy versus digital psychotherapy options for depression: survey of adults in the U.S. NPJ Digit Med. 2019 Feb 11;2:6. doi: 10.1038/s41746-019-0077-1. eCollection 2019. PMID 31304356
- [Background] Andersson G, Titov N, Dear BF, Rozental A, Carlbring P. Internet-delivered psychological treatments: from innovation to implementation. World Psychiatry. 2019 Feb;18(1):20-28. doi: 10.1002/wps.20610. PMID 30600624
- [Background] Jennings KS, Cheung JH, Britt TW, Goguen KN, Jeffirs SM, Peasley AL, Lee AC. How are perceived stigma, self-stigma, and self-reliance related to treatment-seeking? A three-path model. Psychiatr Rehabil J. 2015 Jun;38(2):109-116. doi: 10.1037/prj0000138. Epub 2015 Apr 6. PMID 25844914
- [Background] Swift JK, Callahan JL, Cooper M, Parkin SR. The impact of accommodating client preference in psychotherapy: A meta-analysis. J Clin Psychol. 2018 Nov;74(11):1924-1937. doi: 10.1002/jclp.22680. Epub 2018 Aug 8. PMID 30091140
- [Background] Dorow M, Lobner M, Pabst A, Stein J, Riedel-Heller SG. Preferences for Depression Treatment Including Internet-Based Interventions: Results From a Large Sample of Primary Care Patients. Front Psychiatry. 2018 May 17;9:181. doi: 10.3389/fpsyt.2018.00181. eCollection 2018. PMID 29867605
- [Background] March S, Day J, Ritchie G, Rowe A, Gough J, Hall T, Yuen CYJ, Donovan CL, Ireland M. Attitudes Toward e-Mental Health Services in a Community Sample of Adults: Online Survey. J Med Internet Res. 2018 Feb 19;20(2):e59. doi: 10.2196/jmir.9109. PMID 29459357
- [Background] Lancsar E, Louviere J. Conducting discrete choice experiments to inform healthcare decision making: a user's guide. Pharmacoeconomics. 2008;26(8):661-77. doi: 10.2165/00019053-200826080-00004. PMID 18620460
- [Background] Lambooij MS, Harmsen IA, Veldwijk J, de Melker H, Mollema L, van Weert YW, de Wit GA. Consistency between stated and revealed preferences: a discrete choice experiment and a behavioural experiment on vaccination behaviour compared. BMC Med Res Methodol. 2015 Mar 12;15:19. doi: 10.1186/s12874-015-0010-5. PMID 25887890
- [Background] Muhlbacher AC, Juhnke C, Beyer AR, Garner S. Patient-Focused Benefit-Risk Analysis to Inform Regulatory Decisions: The European Union Perspective. Value Health. 2016 Sep-Oct;19(6):734-740. doi: 10.1016/j.jval.2016.04.006. Epub 2016 Sep 9. PMID 27712699
- [Background] Sicsic J, Pelletier-Fleury N, Moumjid N. Women's Benefits and Harms Trade-Offs in Breast Cancer Screening: Results from a Discrete-Choice Experiment. Value Health. 2018 Jan;21(1):78-88. doi: 10.1016/j.jval.2017.07.003. Epub 2017 Aug 18. PMID 29304944
- [Background] Quaife M, Eakle R, Cabrera Escobar MA, Vickerman P, Kilbourne-Brook M, Mvundura M, Delany-Moretlwe S, Terris-Prestholt F. Divergent Preferences for HIV Prevention: A Discrete Choice Experiment for Multipurpose HIV Prevention Products in South Africa. Med Decis Making. 2018 Jan;38(1):120-133. doi: 10.1177/0272989X17729376. Epub 2017 Sep 1. PMID 28863752
- [Background] Hazlewood GS, Bombardier C, Tomlinson G, Thorne C, Bykerk VP, Thompson A, Tin D, Marshall DA. Treatment preferences of patients with early rheumatoid arthritis: a discrete-choice experiment. Rheumatology (Oxford). 2016 Nov;55(11):1959-1968. doi: 10.1093/rheumatology/kew280. Epub 2016 Jul 31. PMID 27477807
- [Background] Lokkerbol J, Geomini A, van Voorthuijsen J, van Straten A, Tiemens B, Smit F, Risseeuw A, Hiligsmann M. A discrete-choice experiment to assess treatment modality preferences of patients with depression. J Med Econ. 2019 Feb;22(2):178-186. doi: 10.1080/13696998.2018.1555404. Epub 2018 Dec 22. PMID 30501437
- [Background] Reed Johnson F, Lancsar E, Marshall D, Kilambi V, Muhlbacher A, Regier DA, Bresnahan BW, Kanninen B, Bridges JF. Constructing experimental designs for discrete-choice experiments: report of the ISPOR Conjoint Analysis Experimental Design Good Research Practices Task Force. Value Health. 2013 Jan-Feb;16(1):3-13. doi: 10.1016/j.jval.2012.08.2223. PMID 23337210
- [Background] Veldwijk J, Lambooij MS, de Bekker-Grob EW, Smit HA, de Wit GA. The effect of including an opt-out option in discrete choice experiments. PLoS One. 2014 Nov 3;9(11):e111805. doi: 10.1371/journal.pone.0111805. eCollection 2014. PMID 25365169
- [Background] Tunnessen M, Hiligsmann M, Stock S, Vennedey V. Patients' preferences for the treatment of anxiety and depressive disorders: a systematic review of discrete choice experiments. J Med Econ. 2020 Jun;23(6):546-556. doi: 10.1080/13696998.2020.1725022. Epub 2020 Feb 24. PMID 32011209
- [Background] de Bekker-Grob EW, Donkers B, Jonker MF, Stolk EA. Sample Size Requirements for Discrete-Choice Experiments in Healthcare: a Practical Guide. Patient. 2015 Oct;8(5):373-84. doi: 10.1007/s40271-015-0118-z. PMID 25726010
- [Background] Marshall D, Bridges JF, Hauber B, Cameron R, Donnalley L, Fyie K, Johnson FR. Conjoint Analysis Applications in Health - How are Studies being Designed and Reported?: An Update on Current Practice in the Published Literature between 2005 and 2008. Patient. 2010 Dec 1;3(4):249-56. doi: 10.2165/11539650-000000000-00000. PMID 22273432
- [Background] Noble H, Smith J. Issues of validity and reliability in qualitative research. Evid Based Nurs. 2015 Apr;18(2):34-5. doi: 10.1136/eb-2015-102054. Epub 2015 Feb 4. No abstract available. PMID 25653237
- [Background] Leigh S, Ashall-Payne L, Andrews T. Barriers and Facilitators to the Adoption of Mobile Health Among Health Care Professionals From the United Kingdom: Discrete Choice Experiment. JMIR Mhealth Uhealth. 2020 Jul 6;8(7):e17704. doi: 10.2196/17704. PMID 32628118
- [Background] McGrady ME, Pai ALH, Prosser LA. Using discrete choice experiments to develop and deliver patient-centered psychological interventions: a systematic review. Health Psychol Rev. 2021 Jun;15(2):314-332. doi: 10.1080/17437199.2020.1715813. Epub 2020 Jan 22. PMID 31937184
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941